CLINICAL TRIAL: NCT01662505
Title: An Open Label, Phase I Trial of Intravenous Once Every 2 Weeks Administration of BI 6727 (Volasertib) in Japanese Patients With Acute Myeloid Leukemia
Brief Title: Volasertib in Japanese Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.26
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BI 6727

ARMS (1):
- Volasertib (Experimental): Patient to receive escalating dose of volasertib
  Interventions: Drug: Volasertib

INTERVENTIONS:
Drug: Volasertib — Patient to receive volasertib

SUMMARY:
To investigate safety, tolerability, maximum tolerated dose of volasertib in Japanese patients with AML

ELIGIBILITY:
Inclusion criteria:

1. Patients with diagnosis of AML (except for acute promyelocytic leukemia, APL) according to the World Health Organization definition and with one of the following features at screening

   * Relapsed or refractory AML
   * Untreated AML patients not considered to be suitable for standard induction therapy according to investigator's judgement
2. Male or female patients of age >/= 18 years at the time of informed consent
3. Eastern Cooperative Oncology Group performance status score 0 - 2 at screening
4. Signed written informed consent consistent with Japanese Good Clinical Practice.

Exclusion criteria:

1. Patients with APL
2. Patients in the third or later relapse
3. Prior stem cell transplantation
4. Treatment with systemic therapy for the primary disease (including an investigational drug) within 14 days before the first dose of volasertib with the exception of hydroxyurea, or lack of recovery from any acute toxicities or clinically significant adverse events pertinent to the prior systemic therapy
5. Treatment with gemtuzumab ozogamicin within 6 weeks before the first dose of volasertib
6. Concomitant medication/treatment with anti-leukemic chemotherapy (systemic or intrathecal), radiotherapy, immunotherapy, or any investigational agent while receiving study treatment
7. Other malignancy requiring treatment at the time of screening
8. Clinical central nervous system (CNS) symptoms deemed by the investigator to be related to leukemic CNS involvement or requiring treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- Japan (6):
  - Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Isehara, Kanagawa
  - Boehringer Ingelheim Investigational Site, Maebashi, Gunma,
  - Boehringer Ingelheim Investigational Site, Nagasaki, Nagasaki
  - Boehringer Ingelheim Investigational Site, Nagoya-shi, Aichi
  - Boehringer Ingelheim Investigational Site, Yoshida-gun, Fukui

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with written informed consent underwent screening within (≤) 14 days before starting the volasertib treatment. Eligible patients were enrolled and treated as soon as possible or within (≤)14 days after obtaining informed consent.
Groups:
- V 350 mg: Patients received 350 milligram (mg) of volasertib (V) as monotherapy on Days 1 and 15 of a 28-day cycle via intravenous (i.v.) drip infusion over 2 hours.
- V 400 mg: Patients received 400 mg of volasertib as monotherapy on Days 1 and 15 of a 28-day cycle via i.v. drip infusion over 2 hours.
- V 450 mg: Patients received 450 mg of volasertib as monotherapy on Days 1 and 15 of a 28-day cycle via i.v. drip infusion over 2 hours.
Period: Overall Study
Arm/Group | V 350 mg | V 400 mg | V 450 mg
Started | 7 | 4 | 8
Completed | 0 | 0 | 0
Not Completed | 7 | 4 | 8
Not completed — Progressive disease | 6 | 1 | 5
Not completed — Refused cont. medication | 0 | 0 | 1
Not completed — Not specified above | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients that received at least 1 dose of the trial medication were defined as the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | V 350 mg | V 400 mg | V 450 mg | Total
Number analyzed (Participants) | 7 | 4 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.4 (6.0) | 78.0 (5.9) | 69.1 (8.6) | 72.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) in Cycle 1 for the Determination of the Maximum Tolerated Dose (MTD) of Volasertib
Description: Primary objective for this trial was to identify the MTD of volasertib. The MTD was defined as the highest dose level at which DLTs were reported in at most 2 in 6 evaluable patients during cycle 1. In this outcome measure the number of participants with DLTs in cycle 1 is presented.
Time Frame: From first administration of trial drug up to 28 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | V 350 mg | V 400 mg | V 450 mg
Number analyzed (Participants) | 7 | 4 | 8
Participants | 0 | 0 | 1

2. Secondary Outcome: Best Response by Complete Remission (CR)
Description: The secondary outcome best response will be presented by the CR, CR with incomplete blood count recovery (CRi) and partial remission (PR).
  In this outcome measure the CR will be presented.
  The criteria for the CR are:
  Bone marrow blasts less than 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) >1.0 × 10^9/Litre (L) (1000/microlitre (μL)); platelet count >100 × 10^9/L (100 000/μL); independence of red cell transfusions.
Time Frame: From first administration of trial drug up to 486 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | V 350 mg | V 400 mg | V 450 mg
Number analyzed (Participants) | 7 | 4 | 8
Participants | 1 | 0 | 2

3. Primary Outcome: MTD of Volasertib
Description: Primary objective for this trial was to identify the MTD of volasertib. The MTD was defined as the highest dose level at which DLTs were reported in at most 2 in 6 evaluable patients during cycle 1. In this outcome measure the MTD is presented.
Time Frame: From first administration of trial drug up to 28 days
Population: Treated Set
Measure: Number; unit: milligram (mg)
Groups:
- Volasertib: Patients received volasertib as monotherapy on Days 1 and 15 of a 28-day cycle via i.v. drip infusion over 2 hours.
Arm/Group | Volasertib
Number analyzed (Participants) | 8
milligram (mg) | 450

4. Secondary Outcome: Best Response by CRi
Description: The secondary outcome best response will be presented by the CR, CRi and PR. In this outcome measure the CRi will be presented.
  The criteria for the CRi are:
  All CR criteria are met except for residual neutropenia (<1.0 × 10^9/L [1000/μL]) or thrombocytopenia (<100 × 10^9/L [100 000/μL]).
Time Frame: From first administration of trial drug up to 486 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | V 350 mg | V 400 mg | V 450 mg
Number analyzed (Participants) | 7 | 4 | 8
Participants | 0 | 2 | 1

5. Secondary Outcome: Best Response by PR
Description: The secondary outcome best response will be presented by the CR, CRi and PR. In this outcome measure the PR is presented.
  The criteria for the PR are:
  All haematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Time Frame: From first administration of trial drug up to 486 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | V 350 mg | V 400 mg | V 450 mg
Number analyzed (Participants) | 7 | 4 | 8
Participants | 0 | 0 | 1

6. Secondary Outcome: Remission Duration
Description: The remission duration is the time from the date of achieving CR or CRi until relapse for patients with documented CR or CRi.
Time Frame: From first administration of trial drug up to 486 days
Population: Treated Set, patient with remissions
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | V 350 mg | V 400 mg | V 450 mg
Number analyzed (Participants) | 1 | 2 | 3
Days | 358.0 (NA) — N=1 | 72.0 (2.8) | 170.3 (164.6)

ADVERSE EVENTS:
Time Frame: From inclusion into the study to 21 days after last drug administration (up to 507 days)
Arm/Group | V 350 mg | V 400 mg | V 450 mg
Serious Adverse Events (participants affected / at risk) | 3/7 | 0/4 | 4/8
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V 350 mg (N=7) | V 400 mg (N=4) | V 450 mg (N=8)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V 350 mg (N=7) | V 400 mg (N=4) | V 450 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 6
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 0
Cheilosis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1 | 1
Lip erosion (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 4
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Catheter site erosion (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 1
Injection site reaction (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 2
Soft tissue inflammation (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0
Bacillus bacteraemia (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
Sepsis (Infections and infestations) | 0 | 1 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urethritis (Infections and infestations) | 0 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time abnormal (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
International normalised ratio (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1
Vascular pain (Vascular disorders) | 0 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.